CLINICAL TRIAL: NCT06327932
Title: A Multicenter Prospective Randomized Controlled Clinical Trial of Hyperthermic Intravesical Chemotherapy After Transurethral Resection of Bladder Tumors in Patients With Non-Muscle-Invasive Bladder Cancer
Brief Title: HIVEC in Patients With Non-Muscle-Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIVEC(PRG)
Record Dates: First submitted 2024-03-07; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Non-Muscle-Invasive Bladder Cancer
Keywords: Non-Muscle-Invasive Bladder Cancer; Hyperthermic Intravesical Chemotherapy; recurrence rate
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Matched control (Active Comparator): Patients undergo Transurethral Resection of Bladder Tumors (TURBT) and receive Intravesical Chemotherapy.
  Interventions: Procedure: TURBT; Procedure: Intravesical Chemotherapy; Drug: Gemcitabine
- HIVEC (Experimental): Patients undergo Transurethral Resection of Bladder Tumors (TURBT) and Hyperthermic Intravesical Chemotherapy (HIVEC)
  Interventions: Procedure: TURBT; Procedure: HIVEC; Drug: Gemcitabine

INTERVENTIONS:
Procedure: TURBT — Transurethral Resection of Bladder Tumors
Procedure: HIVEC — Hyperthermic Intravesical Chemotherapy with Gemcitabine (3g/150ml NS) at 45 °C for 60 minutes. Induction perfusion was required to start within 4 weeks, once a week (±5 days) for 6 to 8 times. After the last induction infusion, maintenance infusion was performed, once every month (±2 weeks) for 1 year from the first induction infusion.
  Arms: HIVEC
Procedure: Intravesical Chemotherapy — Intravesical Chemotherapy with Gemcitabine (3g/150ml NS). Induction perfusion was required to start within 4 weeks, once a week (±5 days) for 6 to 8 times. After the last induction infusion, maintenance infusion was performed, once every month (±2 weeks) for 1 year from the first induction infusion.
  Arms: Matched control
Drug: Gemcitabine — Gemcitabine (3g/150ml NS).

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Hyperthermic Intravesical Chemotherapy (HIVEC) with Gemcitabine (GEM) after Transurethral Resection of Bladder Tumors (TURBT) in the treatment of medium or high-risk group Non-Muscle-Invasive Bladder Cancer (NMIBC).

DETAILED DESCRIPTION:
In this study, patients with Non-Muscle-Invasive Bladder Cancer (NMIBC) and planed to undergo Transurethral Resection of Bladder Tumors (TURBT) are randomized into HIVEC group and control group. In HIVEC group, HIVEC is performed with Gemcitabine Gemcitabine (3g/150ml NS) at 45 °C for 60 minutes within 4 weeks, once a week (±5 days) for 6 to 8 times, once a month to 1 year. For the patients in the control group, Intravesical Chemotherapy is administered after TURBT. The primary endpoint is 2-year recurrence rate. Secondary end points include 1-year recurrence rate, recurrence-free survival (RFS) rate, disease free survival (DFS) rate, time to treatment failure (TTF), Success rate of therapeutic operation, Instrument performance evaluation, quality of international prostate symptom score, quality of Urinary Symptoms Distress Score. All efficacy analyses are conducted in the intention-to-treat population. Safety analysis include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who did not receive induction perfusion within 4 weeks after complete resection of bladder tumor with TURBT (Patients who were judged by the investigator to be in need of secondary electrotomy, for the last time).
2. Recurrence risk and prognosis of Non-Muscle-Invasive Bladder Cancer were divided into medium-risk group or high-risk group (patients who underwent multiple electrosurgical biopsies, and the pathological results were based on higher grade tumors).
3. KPS score ≥80, expected survival > 30 months.
4. Pathological suggested non-myoinvasive urothelial carcinoma of the bladder.
5. Age between 18 and 70 years, all genders.
6. Volunteer to participate in this clinical trial and written informed consent.

Exclusion Criteria:

1. Patients with bladder cancer in situ.
2. Combined with proven upper urinary tract or urethral tumors.
3. The patients were complicated with bladder perforation, gross hematuria or urinary tract infection of grade 3-4.
4. Patients with urethral discontinuity, urethral stricture, or inability to use a three lumen catheter normally affect perfusion therapy.
5. Patients who had undergone partial cystectomy or abnormal bladder structure were judged by the investigator to be unsuitable for perfusion therapy.
6. Patients with severe coagulation dysfunction.
7. A history of allergy to injected drugs (gemcitabine).
8. History of pelvic radiation, systemic chemotherapy, or immunotherapy.
9. Complicated with cardiovascular, cerebrovascular, hematopoietic, immune system and other serious diseases.
10. Patients with mental illness, substance abuse, alcoholism, and inability to cooperate.
11. Breastfeeding, pregnant, or planning to have a baby in the near future.
12. Recurrent patients with a prior history of BCG or bladder thermoperfusion therapy.
13. Participated in other clinical trials 1 month before the trial.
14. Vesicoureteral regurgitation.
15. The investigator considered it inappropriate to participate in this clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2-year
  The patients were observed for 2 years since they received HIVEC or intravesical chemotherapy，and cystoscopy was repeated every 3 months. If a new tumor-like organism is seen under the microscope, and pathology indicates urothelial carcinoma of the bladder after TURBT or cystoscopic biopsy, the tumor is considered to have recurred. 2-year recurrence rate = number of recurrence cases within 2 years / total number of enrolled cases * 100%.

SECONDARY OUTCOMES:
1-year recurrence rate | 1-year
  1-year recurrence rate = number of recurrence cases within 1 years / total number of enrolled cases * 100%.
Recurrence-free survival (RFS) rate | 2-year
  Recurrence free survival is calculated from the date of randomization to the date of record recurrence or death from any cause, whichever occurred first.
Time to treatment failure | 2-year
  Time to treatment failure is calculated from the date of randomization to the date of treatment discontinuation/termination, including any reason for discontinuation/termination, such as disease progression, death, withdrawal due to adverse events, subject's refusal to continue the study, or use of a new treatment.
Success rate of therapeutic operation | 2-year
  Success rate of therapeutic operation
Quality of international prostate symptom score | Evaluation was performed during the screening period and at 3, 12 and 24 months after initiation of treatment.
  IPSS is International Prostate Symptom Score (IPSS), 0~35, the higher the score, the worse the symptom severity is.
Quality of bother of score | Evaluation was performed during the screening period and at 3, 12 and 24 months after initiation of treatment
  BS is Bother of Score (BS), 0~6, the higher the score, the worse the performance is.BS is the Bother of Score (BS), 0~6, the higher the score, the worse the performance is.

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Cui, MD, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University